CLINICAL TRIAL: NCT02403453
Title: RHINE™ Cervical Disc Clinical Study
Brief Title: RHINE™ Cervical Disc Clinical Study: A Prospective Observational Study for Patients Requiring 1-2 Level C-spine Surgery
Status: Terminated | Type: Observational
Why Stopped: Stryker has made the decision to remove the Rhine Cervical Disc Replacement from their product portfolio. Stryker is not aware of any safety or effectiveness concerns and this decision is not related to poor patient outcomes or known device failures.
Sponsor: K2M, Inc. (Industry)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-009
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Radiculopathy; Myelopathy; Spondylosis; Herniated Nucleus Pulposus
Keywords: Radiculopathy; Myelopathy; Spondylosis; Herniated Nucleus Pulposus; C3-C7; Osteophytes; Neurological deficit
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases; Spondylosis; Osteophyte; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Rhine Cervical Disc — RHINE Cervical Disc

SUMMARY:
A Prospective, open label, multi-center observational study of patients requiring surgical treatment at one or two (contiguous) cervical spine levels. The primary objectives of the RHINE Cervical Disc study are to: obtain operative data and feedback on surgical instruments and surgical technique; confirm device performance in terms of clinical and radiographic outcomes; confirm device performance in terms of safety and to collect original data to be compared to published reports of the performance of comparable motion-sparing devices, as well as clinical outcomes of fusion devices.

DETAILED DESCRIPTION:
A Prospective, open label, multi-center observational study of patients requiring surgical treatment at one or two (contiguous) cervical spine levels ( C3-C7). The primary objectives of the RHINE Cervical Disc study are to: obtain operative data and feedback on surgical instruments and surgical technique; confirm device performance in terms of clinical and radiographic outcomes; confirm device performance in terms of safety and to collect original data to be compared to published reports of the performance of comparable motion-sparing devices, as well as clinical outcomes of fusion devices. Device- and procedure-related adverse events, serious adverse events, and secondary surgeries will be monitored throughout. AEs will be characterized by severity, seriousness and relationship to device. Investigator reports of serious adverse events and any AE trends will be reviewed by a medical monitor.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires reconstruction of the disc from C3 to C7 following discectomy at 1 or 2 (contiguous) levels for intractable radiculopathy (arm pain and/or a neurological deficit) with or without neck pain, or myelopathy due to abnormality localized to the level of the disc space and at least one of the following conditions confirmed by radiographic imaging (CT, MRI, X-rays): herniated nucleus pulposus, spondylosis (defined by the presence of osteophytes), and/or visible loss of disc height compared to adjacent levels.
* The patient has failed at least 6 weeks of non-operative treatment or demonstrated progressive signs or symptoms despite non-operative treatment prior to implantation.
* Self-reports a pre-operative upper extremity (right or left) VAS pain score ≥ 20 (0-100).
* Self-reports pre-operative NDI score ≥ 30% (raw score of ≥ 15/50).
* Willing and able to comply with the protocol requirements including follow-up visit schedule.
* Willing and able to sign a study specific informed consent.

Exclusion Criteria:

* More than two cervical levels requiring surgery, or has two levels requiring surgery that are not adjacent.
* Previous surgical intervention at the target level(s)
* Any of the following at the target level(s):
* Significant cervical anatomical deformity, e.g., ankylosing spondylitis, rheumatoid arthritis, etc.
* Moderate to advanced spondylosis. Patients who demonstrate advanced degenerative changes characterized by any of the following: bridging osteophytes, marked reduction or absence of motion (< 2 degrees change from flexion to extension), collapse of the intervertebral disc space of greater than 50% of its normal height (compared to adjacent levels)
* Radiographic signs of subluxation > 3.5 mm
* Angulation of the disc space more than 11 degrees greater than adjacent segments
* Significant kyphotic deformity (> 5 degrees) at a single level or significant reversal of lordosis (not corrected with extension)
* Fused level adjacent to a level to be treated
* Axial neck pain is the patient's solitary symptom
* Severe pathology of the facet joints of the involved vertebral bodies
* Previous diagnosis of osteopenia or osteomalacia
* Has any of the following risk factors that may be associated with a diagnosis of osteoporosis.
* Spinal metastases
* Extreme obesity (BMI ≥ 40)
* Overt or active bacterial infection, either local or systemic
* Severe insulin dependent diabetes
* Chronic or acute renal failure or prior history of renal disease
* Fever (temp > 38.3° C oral) at the time of surgery
* Documented allergy or intolerance to titanium or polyurethane
* Reported concomitant conditions requiring daily, high-dose oral and/or inhaled steroids.
* Any medical condition that may interfere with the postoperative management program or preclude meaningful patient self-assessments, e.g., advanced emphysema, progressive neurological disease, or Alzheimer's disease
* Any medical condition that may result in patient death prior to study completion, e.g., unstable cardiac disease, active malignancy
* History of an endocrine or metabolic disorder known to affect osteogenesis
* Active immunosuppressive disorder that may predispose patient to infection
* Participating in or planning to participate in another clinical study that might influence the treatment outcomes or ability to comply with the study requirements
* Member of a vulnerable population such as, mentally incompetent, prisoner
* Pregnant, nursing, considering becoming pregnant during the study, or is of childbearing potential and unwilling to use an accepted form of birth control during the study.
* History or suspicion of substance abuse or currently undergoing substance abuse treatment
* In the judgment of the Investigator, patient is not likely to be able to fulfill the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for the study enrollment will be skeletally mature patients undergoing reconstruction of the disc from C3 to C7 following discectomy at one or two contiguous levels for intractable radiculopathy (arm pain and/or a neurological deficit) with or without neck pain, or myelopathy due to abnormality localized to the level of the disc space and at least one of the following conditions confirmed by radiographic imaging (CT, MRI, X-rays): herniated nucleus pulposus, spondylosis (defined by the presence of osteophytes), and/or visible loss of disc height compared to adjacent levels. Patients should have failed at least 6 weeks of non-operative treatment or demonstrated progressive signs or symptoms despite non-operative treatment prior to implantation.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) change from baseline | Pre-operative, 6 months, 12 months, 24 months and 60 months
  Evaluation of the change in function will be scored using the Neck Disability Index (NDI) at all time points compared to baseline (pre-operative). NDI is a subject-completed, condition-specific functional status questionnaire with 10 questions. Each question is scored from 0 to 5, summed to a total and multiplied by 2 to get a score from 0 to 100. A 15 point change in NDI score compared with baseline (pre-operative score) will be used as the measure for a clinically significant change.
Radiographic Outcomes | Pre-operative, 6-12 weeks, 6 months, 12 months, 24 months and 60 months
  Anteroposterior & Lateral ( or MRI at Pre-operative ) and Flexion and Extension x-rays will be taken at all time points. An independent radiologist will review and assess all radiographs including: range of motion, translation, intervertebral height, device height, device positioning/migration, heterotopic ossification and adjacent segment degeneration.
Number of Patients with Adverse Events (AEs) | Up to 6-12 weeks post-discharge , 6 months, 12 months, 24 months annd 60 months
  AEs will be monitored throughout the study and characterized by seriousness, severity and relationship to the device and procedure, at a minimum.

SECONDARY OUTCOMES:
Pain: Neck, Right Arm, Left Arm, Worst arm Visual analog Scale Change form Baseline | Pre-operative, 6-12 weeks post-discharge , 6 months, 12 months, 24 months annd 60 months
  The intensity of neck pain, right arm pain and left arm pain will be evaluated using a 100 mm VAS. The scale is measured from 0 mm (no pain) to 100 mm (extreme pain). The VAS will be scored at all time points and compared to baseline (pre-operative). A change of 15 mm is considered clinically significant.
Secondary Surgeries (Surgical Interventions) | Up to 6-12 weeks post-discharge , 6 months, 12 months, 24 months and 60 months
  Secondary surgeries will be described and will be classified as follows:
  * Index Level Revision without Implant Removal: a procedure that adjusts or in any way modifies the original implant configuration without removal of the original implant, e.g., adjusting the position of the implant, or adding supplemental fixation.
  * Index Level Revision with Implant Removal: a procedure that removes the original implant, with replacement using a new implant or without replacement.
  * Adjacent Level Surgery: any surgical procedure at a level adjacent to the treated level(s) that does not remove, modify or add any components to the implant configuration.
  * Other Spine Surgery: surgery at spine level that is not an index or adjacent level.
  Surgeries unrelated to the spine will not be recorded as secondary surgeries but the adverse effect leading to the surgery will be recorded on an AE form and characterized as an 'inpatient hospitalization.
Quality of life (SF-36) | Pre-operative, 6 months, 12 months, 24 months annd 60 months
  SF-36 survey will be used to calculate overall, mental (MCS) and physical (PCS) component scores at all post-op time-points compared to baseline (pre-operative)
Functional / Economic Impact - Prolo Scale | Pre-operative, 6 months, 12 months, 24 months annd 60 months
  It is a 10-point scale consisting of only 2 questions evaluating the functional and economic status of patients. Scores 9-10 are considered excellent , scores less than 4 are considered poor.
Neurological function | Pre-operative, 6 months, 12 months, 24 months annd 60 months
  Neurological function will be assessed pre-operatively and all post-op visits, unscheduled visits to assess an Adverse Event, by evaluating:
  * Reflexes (0-4)
  * Signs of myelopathy (Hoffman's, Babinski, Ankle Clonus)
  * Sensory (light touch, pin prick; impaired/normal)
  * Motor strength (0-5)
  Maintenance or improvement in neurological function for this study is defined as: No clinically significant worsening at any post-operative time point that is permanent (compared to baseline or best neurological result post-operatively)
Global Assessment | 6 months, 12 months, 24 months and 60 months
  Subject's self-reported assessment of improvement in their neck/arm problem since treatment. Scored on a 4-pt scale (much better, better, unchanged, worse) at 6, 12, 24 and 60 months.
Patient satisfaction | 6 months, 12 months, 24 months and 60 months
  This will be based on subject's self-reported response to whether he/she is satisfied with the outcome of his/her neck surgery, scored on a 4-pt scale (strongly agrees, agrees, disagrees, strongly disagrees) at 6, 12, 24 and 60 months.
Patient treatment success (PTS) | 24 months
  Patients should have met all the of the following criteria:
  * ≥ 15 point improvement in NDI compared to baseline (pre-operative),
  * No new or increased permanent, clinically significant neurological deficit compared to baseline (pre-operative),
  * No device-related surgical intervention (specifically, intra-operative serious device-related AEs (implant or instrument) or conversion to fusion, or device-related secondary surgery at index level).
Use of NSAIDS and other pain Medications. | Pre-operative, 6 months, 12 months, 24 months annd 60 months
  Will document duration of prescribed post-operative use of NSAIDS (≤2 weeks, >2 weeks), and use (frequency and potency) of medications to manage c-spine condition at each follow-up interval compared with pre-operative level of management.
Estimated blood loss | During Operation
  The amount of blood loss over the entire length of the surgery, documented on the Anesthesia Record, will be captured.
Surgery time | During Operation
  The length of surgical procedure from the initial incision to final closure will be captured from the Anesthesia Record.
Length of hospital stay | At discharge, estimated average of 3-6 days after surgery
  The length of hospital stay from date of admission to date of discharge will be calculated.
Surgeon satisfaction with instruments and surgical technique | At discharge, estimated average of 3-6 days after surgery
  4-pt scale (very satisfied, satisfied, somewhat unsatisfied, very unsatisfied)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Hagg O, Fritzell P, Oden A, Nordwall A; Swedish Lumbar Spine Study Group. Simplifying outcome measurement: evaluation of instruments for measuring outcome after fusion surgery for chronic low back pain. Spine (Phila Pa 1976). 2002 Jun 1;27(11):1213-22. doi: 10.1097/00007632-200206010-00014. PMID 12045520
- [Background] Mehren C, Suchomel P, Grochulla F, Barsa P, Sourkova P, Hradil J, Korge A, Mayer HM. Heterotopic ossification in total cervical artificial disc replacement. Spine (Phila Pa 1976). 2006 Nov 15;31(24):2802-6. doi: 10.1097/01.brs.0000245852.70594.d5. PMID 17108833
- [Background] McAfee PC, Cunningham BW, Devine J, Williams E, Yu-Yahiro J. Classification of heterotopic ossification (HO) in artificial disk replacement. J Spinal Disord Tech. 2003 Aug;16(4):384-9. doi: 10.1097/00024720-200308000-00010. PMID 12902954
- [Background] Beaurain J, Bernard P, Dufour T, Fuentes JM, Hovorka I, Huppert J, Steib JP, Vital JM, Aubourg L, Vila T. Intermediate clinical and radiological results of cervical TDR (Mobi-C) with up to 2 years of follow-up. Eur Spine J. 2009 Jun;18(6):841-50. doi: 10.1007/s00586-009-1017-6. Epub 2009 May 12. PMID 19434431
- [Background] Geisler FH, Blumenthal SL, Guyer RD, McAfee PC, Regan JJ, Johnson JP, Mullin B. Neurological complications of lumbar artificial disc replacement and comparison of clinical results with those related to lumbar arthrodesis in the literature: results of a multicenter, prospective, randomized investigational device exemption study of Charite intervertebral disc. Invited submission from the Joint Section Meeting on Disorders of the Spine and Peripheral Nerves, March 2004. J Neurosurg Spine. 2004 Sep;1(2):143-54. doi: 10.3171/spi.2004.1.2.0143. PMID 15346999